CLINICAL TRIAL: NCT05728879
Title: Characterization of the Microbiome in Cutaneous T Cell Lymphoma Skin Lesions Before and After Use of APR-TD011® (RLF-TD011®) Spray Solution
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Xiaolong (Alan) Zhou, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00217913
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cutaneous T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CTCL participants (Experimental): Visits will include screening, pre-treatment (week 0), weeks 4 and 8.
  Interventions: Combination Product: APR-TD011 (RLF-TD011)

INTERVENTIONS:
Combination Product: APR-TD011 (RLF-TD011) — APR-TD011 (RLF-TD011) wound cleansing spray (drug/device combination product with a 510k clearance that is commercially marketed in the US for use by or on the order of a physician.
  Other Names: Nexodyn AOS

SUMMARY:
This open-label, pilot study will evaluate the tolerance and change in the microbiome from the use of APR-TD011 ((RLF-TD011) wound cleansing spray for the treatment of CTCL skin lesions.

ELIGIBILITY:
Inclusion Criteria:

* Adults with early-stage mycosis fungoides (stages IA-IB)
* At least two target lesions that have been present for at least 3 weeks and is at least 10 cm2 , so that at least one lesion may be allocated to each of the treatment regimes
* Target lesion with swab that is culture positive for staphylococcus aureus, but not to an extent that would require systemic antibiotics
* Agree to avoid washing or using a topical application at the target lesion starting the night before each scheduled study visit.
* Agree for the duration of study participation to avoid using dilute bleach or vinegar baths, or other antiseptic use, at the target lesion from screening throughout the study.

Exclusion Criteria:

* Patients currently or recently (within past 4 weeks) on topical or systemic antibiotics adults unable to provide informed consent, (infants, children, teenagers, pregnant women, prisoners and other vulnerable populations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in microbiome species | 4 weeks
  Reduction of Staphylococcus aureus relative abundance between baseline and Week 4

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology CTU, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No